CLINICAL TRIAL: NCT02733588
Title: A Phase 2 Proof-of-Concept Study of Sensor-Guided, Clinician-Administered Delivery of G-Pump™ (Glucagon Infusion) From an OmniPod® to Prevent Post-Prandial Hypoglycemia in Post-Bariatric Surgery Patients
Brief Title: Delivery of G-Pump™ (Glucagon Infusion) From an OmniPod® to Prevent Hypoglycemia in Post-Bariatric Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XSGO-PB01; 1R44DK107114-01 (NIH)
Record Dates: First submitted 2016-03-30; First posted 2016-04-11 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Hypoglycemia; Complications of Bariatric Procedures
Keywords: hypoglycemia; glucagon; glucose metabolism disorders; hormones; gastrointestinal agents; bariatric surgery; incretins
MeSH Terms: conditions — Hypoglycemia; Glucose Metabolism Disorders | interventions — Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- G-Pump™ (glucagon infusion) (Experimental): 0.15 or 0.3 mg G-Pump™ (glucagon infusion) administered from OmniPod® pump
  Interventions: Drug: G-Pump™ (glucagon infusion)

INTERVENTIONS:
Drug: G-Pump™ (glucagon infusion) — 0.15 or 0.3 mg G-Pump™ (glucagon infusion) administered from OmniPod® pump
  Other Names: glucagon

SUMMARY:
The primary objective of this study is to test an optimized control system for sensor-guided (physician administered) delivery of glucagon, and test Proof-of-Concept (POC) in a clinical setting in patients with severe hypoglycemia following bariatric surgery.

DETAILED DESCRIPTION:
This is a Phase 2a, single-center, open-label, proof-of-concept study designed to test the ability of the control algorithm to detect and direct timing of G-Pump™ glucagon infused from an OmniPod® pump to prevent hypoglycemia in patients with post-bariatric hypoglycemia syndrome. While the algorithm will provide an alert as to when glucagon should be dosed to prevent hypoglycemia, there will be no automation in this clinical trial and it will ultimately be up to the physician to initiate dosing via the OmniPod® controller.

Participant on continuous glucose monitoring will arrive at the clinic and IV line will be inserted for venous access. Subject will then be asked to drink a liquid mixed meal containing 60 g of carbohydrates, e.g. Boost® Nutritional Drink, over 10 minutes. Blood samples will be collected for glucose and hormone measurement.

The open-loop system will be set to recognize low sensor glucose values, triggering an alert to the physician, who will deliver a bolus of 150 or 300 µg of glucagon via the pump, with the goal of preventing further decline in glucose values. Depending on response, a second bolus dose of 150 or 300 µg of glucagon may be administered. Plasma glucose will be measured after glucagon administration to ensure successful treatment and glucose stability, and glucagon levels will be analyzed concurrently to determine magnitude of increase above baseline. Sensors will be downloaded for subsequent analysis of appropriateness of alert timing and trigger for glucagon bolus delivery.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with ongoing post-bariatric hypoglycemia with prior episodes of neuroglycopenia, unresponsive to dietary intervention (low glycemic index, controlled carbohydrate portions) and trial of acarbose therapy at the maximally tolerated dose.
* willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.

Exclusion Criteria:

* documented hypoglycemia occurring in the fasting state (> 12 hours fast);
* chronic kidney disease stage 4 or 5;
* hepatic disease, including serum alanine aminotransferase or aspartate aminotransferase greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
* congestive heart failure, New York Heart Association class II, III or IV;
* history of myocardial infarction, unstable angina or revascularization within the past 6 months;
* history of a cerebrovascular accident;
* seizure disorder (other than with suspect or documented hypoglycemia);
* active treatment with any diabetes medications except for acarbose;
* active malignancy, except basal cell or squamous cell skin cancers;
* personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease);
* known insulinoma;
* major surgical operation within 30 days prior to screening;
* hematocrit ≤ 33%;
* bleeding disorder, treatment with warfarin, or platelet count <50,000;
* blood donation (1 pint of whole blood) within the past 2 months;
* active alcohol abuse or substance abuse;
* current administration of oral or parenteral corticosteroids;
* pregnancy and/ or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study.
* use of an investigational drug within 30 days prior to screening.
* there will be no involvement of special vulnerable populations such as pregnant women, prisoners, institutionalized or incarcerated individuals, or others who may be considered vulnerable populations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04-05 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laguna Sanz AJ, Mulla CM, Fowler KM, Cloutier E, Goldfine AB, Newswanger B, Cummins M, Deshpande S, Prestrelski SJ, Strange P, Zisser H, Doyle FJ 3rd, Dassau E, Patti ME. Design and Clinical Evaluation of a Novel Low-Glucose Prediction Algorithm with Mini-Dose Stable Glucagon Delivery in Post-Bariatric Hypoglycemia. Diabetes Technol Ther. 2018 Feb;20(2):127-139. doi: 10.1089/dia.2017.0298. PMID 29355439

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 8 patients were enrolled in the study. One subject withdrew prior to completing study procedures, leaving 7 subjects who were assigned to a treatment arm. Consistent with the number of subjects who started treatment period 1, the number enrolled is given as 7 even though demographics are presented for all 8 qualified/enrolled subjects.
Period: Overall Study
Arm/Group | G-Pump™ (Glucagon Infusion)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 8 subjects were enrolled into the study and demographic characteristics are provided for these 8 subjects. One subject dropped out before receiving study treatment or beginning any study procedures. A total of 7 unique subjects received treatment, and due to the iterative nature of the study, 2 subjects participated twice.
Arm/Group | G-Pump™ (Glucagon Infusion)
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 51 [38 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Months postop hypoglycemia diagnosed [Mean (Full Range); unit: months] | 41 [12 to 150]
Months postop at study visit [Median (Full Range); unit: months] | 116 [45 to 176]
Hemoglobin A1c [Mean (Full Range); unit: %] | 5.7 [5.4 to 5.8]
Preoperative Body Mass Index (BMI) [Mean (Full Range); unit: kg/m2] | 46.4 [37.8 to 61.0]
Current BMI [Mean (Full Range); unit: kg/m2] | 30.1 [24.3 to 36.8]
Delta BMI [Mean (Full Range); unit: kg/m2] | -16.3 [-36.7 to -5.2]
Prescribed glucose-modifying medications [Count of Participants; unit: Participants] | 6
Received nutritional counseling [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Detection/Notification of Hypoglycemia
Description: Frequency with which the device controller software correctly identifies impending hypoglycemia (glucose < 75 mg/dl) and notifies the investigator to initiate treatment. Reported as the number of successful identifications.
Time Frame: 0 - 120 minutes following dosing
Population: Includes all subjects who completed a study visit, including repeat visits by 2 subjects.
Measure: Number; unit: successful events
Arm/Group | G-Pump™ (Glucagon Infusion)
Number analyzed (Participants) | 9
successful events | 9

2. Secondary Outcome: Number of Subjects With Severe Hypoglycemia
Description: Frequency of severe hypoglycemia defined as glucose levels below 60 mg/dl. Reported as the number of subjects with severe hypoglycemia.
Time Frame: 0 - 120 minutes following dosing
Population: Includes all subjects who completed a study visit, including repeat visits by 2 subjects.
Measure: Number; unit: participants
Arm/Group | G-Pump™ (Glucagon Infusion)
Number analyzed (Participants) | 9
participants | 3

3. Secondary Outcome: Number of Subjects With Rebound Hyperglycemia
Description: Frequency of rebound hyperglycemia defined as glucose levels above 180 mg/dl. Reported as the number of subjects with rebound hyperglycemia.
Time Frame: 0 - 120 minutes following dosing
Population: Includes all subjects who completed a study visit, including repeat visits by 2 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pump™ (Glucagon Infusion)
Number analyzed (Participants) | 9
Participants | 0

4. Secondary Outcome: Glucose Time in Range
Description: Time glucose remains in goal range, 60-180 mg/dl, reported in minutes
Time Frame: 0 - 120 minutes following dosing
Population: Includes all subjects who completed a study visit, including repeat visits by 2 subjects.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | G-Pump™ (Glucagon Infusion)
Number analyzed (Participants) | 9
Minutes | 113 (11)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from enrollment until 1 day following the last study visit. Thus the total monitored period was approximately 1 month per patient.
Arm/Group | G-Pump™ (Glucagon Infusion)
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Pump™ (Glucagon Infusion) (N=7)
Nausea (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 2 (2)
Lightheadedness (Nervous system disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Infusion site erythema (Skin and subcutaneous tissue disorders) | 7 (7)
Infusion site edema (Skin and subcutaneous tissue disorders) | 4 (4)
Infusion site discomfort (Skin and subcutaneous tissue disorders) | 4 (4)
Hypoglycemia, post-discharge (Metabolism and nutrition disorders) | 3 (3)
Bleeding from catheter site upon pump removal (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size was small; gender mix, although unequal, is typical of the PBH population at Joslin. The protocol was modified at every stage to test iterations of the detection algorithm and/or increasing glucagon doses to prevent hypoglycemia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT02733588/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT02733588/SAP_001.pdf